CLINICAL TRIAL: NCT01550718
Title: Two Interventions for Early Stage Dementia: A Comparative Efficacy Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Rebecca Logsdon, Research Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 41577-G
Record Dates: First submitted 2012-03-05; First posted 2012-03-12 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Dementia
Keywords: Aerobic Exercise; Alzheimer's Disease; Burden and Stress; Caregiving Issues; Quality of Life; Early Stage Memory Loss
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ESML-Exercise (Physical Activity Program) (Active Comparator): ESML-Exercise consists of four weekly 90-minute classes. Each class includes exercises and a brief discussion of a specific health topic. Classes are carried out in small groups of five to six participant/care partner dyads (10-12 people total), to ensure everyone in the class gets individual attention and that all exercises are done safely using proper form.
  Interventions: Behavioral: ESML-EX (Physical Activity Program)
- ESML-SOCIAL (Social Activity Program) (Active Comparator): ESML-SOCIAL consists of four weekly 90-minute seminars. Each seminar includes discussion of a specific topic, open time for socializing, and a "homework" assignment to be completed prior to the next session. Seminars are carried out in small groups of five to six participant/care partner dyads (10-12 people total), to ensure everyone in the seminar gets individual attention and that everyone has a chance to bring up any concerns.
  Interventions: Behavioral: ESML-Social (Social Activity Program)
- No Intervention (No Intervention): This arm will receive no intervention during the active treatment period. After the 4 month assessment participants can choose to attend a support group.

INTERVENTIONS:
Behavioral: ESML-EX (Physical Activity Program) — ESML-EX consists of four weekly 90-minute classes. Each class includes exercises and a brief discussion of a specific health topic.
  Arms: ESML-Exercise (Physical Activity Program)
Behavioral: ESML-Social (Social Activity Program) — ESML-SOCIAL consists of four weekly 90-minute seminars. Each seminar includes discussion of a specific topic, open time for socializing, and a "homework" assignment to be completed prior to the next session.
  Arms: ESML-SOCIAL (Social Activity Program)

SUMMARY:
Alzheimer's disease (AD) is increasing exponentially, with a projected quadrupling of cases by the mid 21st century. Individuals with AD are at increased risk for a host of medical and psychiatric conditions, and evidence is accumulating supporting the efficacy and effectiveness of psychosocial interventions for improving their mood, function, health, and quality of life. Such interventions are likely to be most effective when they are implemented during the early stages of dementia, when individuals and their family members are coping with the initial diagnosis and associated changes in abilities and activities. Recent randomized clinical trials by the Principal Investigator and colleagues have developed two non-pharmacologic interventions to reduce the social, psychological, physical, and behavioral impact of dementia. This investigation is focused on facilitating their translation into ongoing community-based programs, such as those provided by Alzheimer's Association chapters, senior centers, retirement homes, and other health care providers. The core content of each intervention has been retained in order to maintain or improve their efficacy, and each has been modified to a 4-week group format to increase efficiency of delivery. These modified interventions (ESML-Social and ESML-Ex) will be compared to each other and to a usual care (UC) control group. Outcomes will be assessed at baseline, 1-month post treatment, and 4 month follow-up. Primary outcomes at the 1-month assessment include: social activity participation, family communication, physical activity participation, and physical function. Primary outcomes at 4-month follow up include overall quality of life and depression. It is hypothesized that ESML-Ex and ESML-Social both will have greater improvements than UC. It is hypothesized that ESML-Social will have greater improvements in social participation and family communication than ESML-Ex and UC. It is hypothesized that ESML-Ex will have greater improvements in physical activity participation and physical functioning than ESML-Social and UC. If successful, these 4-week programs may be developed into "modules" that can be incorporated into programming for individuals with early stage dementia in a variety of community settings.

ELIGIBILITY:
Inclusion Criteria:

* Dementia diagnosis
* Clinical Dementia Rating Scale score
* Care Partner agrees to participate with care recipient
* Care recipient lives in the community or a retirement home
* Both care partner and recipient speak English

Exclusion Criteria:

* Significant physical or psychiatric illness in either care partner or care recipient that would prevent participant in a exercise program
* Planning to move out of study area during the 4 month follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Social Activity at post-treatment (1 month) | Baseline and post treatment (1 month)
  The Pleasant Events Schedule-AD, long version, will be used to evaluate social participation and activity.
Change from Baseline in Physical Activity at post-treatment (1 month) | Baseline and post-treatment (1 month)
  The Physical Activity Scale for the Elderly (PASE) will be used to assess level of physical activity of participants and care partners.
Change from Baseline in Quality of Life at post-treatment (1 month) | Baseline and post treatment (1 month)
  The Quality of Life-AD (QOL-AD)scale will measure quality of life domains identified as important for cognitively impaired older adults.
Change from Baseline in Social Activity at 4 month follow-up | Baseline and 4 month follow-up
  The Pleasant Events Schedule-AD, long version, will be used to evaluate social participation and activity.
Change from Baseline in Physical Activity at 4 month follow-up | Baseline and 4 month follow-up
  The Physical Activity Scale for the Elderly (PASE) will be used to assess level of physical activity of participants and care partners.
Change from Baseline in Quality of Life at 4 month follow-up | Baseline and 4 month follow-up
  The Quality of Life-AD (QOL-AD)scale will measure quality of life domains identified as important for cognitively impaired older adults.

SECONDARY OUTCOMES:
Change from Baseline in Communication at post-treatment (1 month) | Baseline and post treatment (1 month)
  The Communication, Affective Expression, and Involvement subscales of the Family Assessment Measure will measure the quality of caregiver-patient communication.
Change from Baseline in Physical Function at post-treatment (1 month) | Baseline and post treatment (1 month)
  The Physical Functioning Scale rates the performance of everyday tasks such as walking around the residence and getting in and out of bed.
Change from Baseline in Mood at post-treatment (1 month) | Baseline and post-treatment (1 month)
  The Geriatric Depression Scale will assess the mood of the participant and their caregiver.
Change from Baseline in Communication at post-treatment (1 month) | Baseline and post-treatment (1 month)
  The Communication, Affective Expression, and Involvement subscales of the Family Assessment Measure will measure the quality of caregiver-patient communication.
Change from Baseline in Physical Functioning at post-treatment (1 month) | Baseline and post-treatment (1 month)
  The Physical Functioning Scale rates the performance of everyday tasks such as walking around the residence and getting in and out of bed.
Change from Baseline in Mood at 4 month follow-up. | Baseline and 4 month follow-up
  The Geriatric Depression Scale will assess the mood of the participant and their caregiver.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca G Logsdon, Ph.D., Principal Investigator — University of Washington
Locations (1):
- UWashington, Seattle, Washington, United States